CLINICAL TRIAL: NCT01441141
Title: Exploratory Studies of Psychophysical Pain Phenotyping and Genetic Variability in Sickle Cell Disease
Brief Title: Genetics and Pain Severity in Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110252; 11-H-0252
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Genotype; Pain; Genetic Variation; Quantitative Sensory Testing (QST); GCH1
Keywords: GCH1; Pain Sensitivity; Quantitative Sensory Testing (QST); Genetic Variation; Sickle Cell Anemia
MeSH Terms: conditions — Pain; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Subjects with SCD
- Arm 2: Subjects without SCD

SUMMARY:
Background:

- Pain is the most common symptom of sickle cell disease. Episodes of severe sickle cell pain are known as "crises." High rates of pain crises are associated with a higher risk of early death. Some people with sickle cell disease have many severe pain crises while others experience fewer crises. This difference in pain crisis may be caused by sensitivity to pain. People with high sensitivity to pain may have more pain crises. Many factors, including a person's genetic makeup, determine sensitivity to pain. Comparing genetic information from people with sickle cell disease and healthy volunteers may provide more information on pain and sickle cell disease.

Objectives:

- To study genetics and pain sensitivity in sickle cell disease.

Eligibility:

* African or African American individuals at least 18 years of age with sickle cell disease.
* Healthy African or African American volunteers at least 18 years of age.

Design:

* Participants will be screened with a medical history and physical exam. They will also provide blood and urine samples.
* Participants will have the following tests:
* Quantitative sensory testing to measure sensitivity to pressure, heat, cold, and mechanical pain.
* EndoPat test to measure blood vessel function and reaction.
* Questionnaires about mood, evidence of depression, pain, quality of sleep, and sleep disturbances.
* Measures of daily pain, whether or not related to sickle cell disease.
* After the first visit, those in the study will have monthly study visits for 6 months. The above tests will be repeated at these visits.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is the most common genetic disease in the United States inherited as an autosomal recessive disorder, where approximately 70,000 individuals have sickle cell disease. Acute painful vaso-occlusive crisis (VOCs) is one of the common complications of SCD that influences overall survival (Platt, Thorington et al. 1991). Pain, is also the most common cause of SCD morbidity, which has a negative impact on quality of life of these individuals and their families. There is significant inter-individual variation in the frequency and course of severe VOCs that result in hospital based treatment, the reasons for which have not been clearly elucidated. Vaso-occlusion of irreversibly sickle red cells within the microcirculation is believed to be the proximate cause of painful VOCs, however it is likely that other non-SCD related factors affecting pain perception and sensitivity to pain will also contribute to individuals susceptibility to pain and therefore contribute to the observed inter-individual variability in the course of VOC. Early identification of individuals who are at high risk for developing severe pain related morbidity and chronic pain syndromes is crucial since early multimodal interventions might have the potential to minimize both the morbidity and mortality associated with VOCs.

<TAB>

Patients with SCD are hypothesized to have lower nitric oxide (NO) bioavailability due to NO scavenging by cell free hemoglobin released into plasma during red cell hemolysis. NO deficiency has been identified as a key factor in development vascular dysfunction in SCD. NO has also recently been identified as a key mediator in processing nociceptive signals and modulation of pain in non-SCD models. Thus, low NO is associated with lower pain perception (Meller, Dykstra et al. 1992; Tegeder, Costigan et al. 2006). GTP cyclohydrolase (GCH1) is the rate-limiting enzyme for synthesis of an essential cofactor for both NO production and metabolism of aromatic amino acids, namely tetrahydrobiopterin (BH4). Therefore it is hypothesized that genetic variants in the GCH1 gene will affect BH4 levels and which will have a secondary impact on vascular dysfunction and sensitivity to pain in SCD.

The primary goal of this protocol is to establish patterns of sensitivity to experimental pain among subjects with SCD compared to healthy African American controls. In addition, an exploratory analysis will determine if increased sensitivity to experimental pain correlates with the frequency and intensity of clinical pain in those with SCD. Once an expected pattern of experimental pain phenotypes are established for a cohort with SCD, we will then further explore the role of GCH1 genetic variants in experimental pain perception and vascular function. If successful, a longer term secondary objective is to establish a sufficiently large patient cohort with experimental pain phenotypes for future exploratory genetic studies to investigate the role of other loci that might influence sensitivity to experimental pain and vascular function in SCD.

ELIGIBILITY:
* ELIGIBILITY CRITERIA FOR ALL PARTICIPANTS:

All study participants must be of self-described African or African American ancestry. They will be at least 18 years old and must be able to provide informed, written consent for participation.

INCLUSION CRITERIA:

Inclusion Criteria for Sickle Cell Patients

1. Diagnosis of sickle cell disease (documentation of SS, SC, S beta + thalassemia, S beta + thalassemia by electrophoresis is required).
2. If taking chronic analgesics (NSAID, acetaminophen) or opioids, study subjects should be on a stable dose for 4 weeks prior to recruitment.

Inclusion Criteria for Control Subjects

1. Hemoglobin AA genotype by HPLC or hemoglobin electrophoresis.
2. General good health defined as the absence of untreated major medical conditions (e.g. uncontrolled systemic hypertension, etc.).

EXCLUSION CRITERIA:

Exclusion Criteria for Sickle Cell Patients

1. History of severe vaso-occlusive pain crisis resulting in either evaluation in an emergency department or admission to a hospital during the two weeks prior to study enrollment.
2. Acute pain at the time of enrollment defined as spontaneous recent onset pain with a self rated score of 6 or higher on a scale of 0-10. (This is acute pain not the pain that subjects function at on a daily basis.)

Exclusion Criteria for Control Subjects

1. Acute pain or injury at enrollment or a recent history of chronic pain (daily pain reported for at least 6 months) in the past 3 years.
2. Major medical/psychiatric illness known to cause pain.
3. Sickle cell trait.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-06-17 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
To determine if thresholds for pain perception are lower in SCD than in non-SCD controls. | Ongoing
  lower pain threshold in SCD than in non-SCD controls

SECONDARY OUTCOMES:
To determine if SCD subjects with higher GCH1 activity have 1) lower pain perception thresholds, 2) a higher prevalence of pain/VOC, 3) altered vascular reactivity and 4) more frequent pain co-morbidities) compared to subjects who lack this. | Ongoing
To determine if variants in the GCH1 gene alter thresholds for pain perception in sickle cell disease. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ataga KI, Moore CG, Jones S, Olajide O, Strayhorn D, Hinderliter A, Orringer EP. Pulmonary hypertension in patients with sickle cell disease: a longitudinal study. Br J Haematol. 2006 Jul;134(1):109-15. doi: 10.1111/j.1365-2141.2006.06110.x. PMID 16803576
- [Background] Bookman EB, Langehorne AA, Eckfeldt JH, Glass KC, Jarvik GP, Klag M, Koski G, Motulsky A, Wilfond B, Manolio TA, Fabsitz RR, Luepker RV; NHLBI Working Group. Reporting genetic results in research studies: summary and recommendations of an NHLBI working group. Am J Med Genet A. 2006 May 15;140(10):1033-40. doi: 10.1002/ajmg.a.31195. PMID 16575896
- [Background] Campbell CM, Kronfli T, Buenaver LF, Smith MT, Berna C, Haythornthwaite JA, Edwards RR. Situational versus dispositional measurement of catastrophizing: associations with pain responses in multiple samples. J Pain. 2010 May;11(5):443-453.e2. doi: 10.1016/j.jpain.2009.08.009. PMID 20439057
- [Derived] Darbari DS, Vaughan KJ, Roskom K, Seamon C, Diaw L, Quinn M, Conrey A, Schechter AN, Haythornthwaite JA, Waclawiw MA, Wallen GR, Belfer I, Taylor JG 6th. Central sensitization associated with low fetal hemoglobin levels in adults with sickle cell anemia. Scand J Pain. 2017 Oct;17:279-286. doi: 10.1016/j.sjpain.2017.08.001. Epub 2017 Sep 30. PMID 28969994
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-H-0252.html